CLINICAL TRIAL: NCT03503695
Title: Auricular Acupuncture for Chronic Pain and Insomnia: a Randomized Clinical Trial
Brief Title: Auricular Acupuncture for Chronic Pain and Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landstuhl Regional Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ann Ketz, Chief, Center for Nursing Science & Clinical Inquiry, Landstuhl Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-10395
Record Dates: First submitted 2018-04-03; First posted 2018-04-20 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Insomnia; Chronic Pain
Keywords: auricular acupuncture; battlefield acupuncture; insomnia; chronic pain; randomized
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular Acupuncture (Active Comparator): Sterile acupuncture semi-permanent (ASP) gold needles will be administered in the following acupuncture points: Cingulate Gyrus, Thalamus point, Omega 2, Point Zero, and Shen Men starting in either ear and alternating left and right until 10 ASP needles are placed. The needles may remain in the AA points for 3-4 days.
  Interventions: Device: Sterile acupuncture semi-permanent (ASP) gold needles
- Comparison Group (No Intervention): There will be no intervention. The participants will be instructed to return on Day 8.

INTERVENTIONS:
Device: Sterile acupuncture semi-permanent (ASP) gold needles
  Other Names: Sedatelac
  Arms: Auricular Acupuncture

SUMMARY:
Background: In the U.S. approximately 1.6 million adults use complementary and alternative or integrative medicine therapy for pain and insomnia. However, very few studies have tested the use of auricular acupuncture (AA) using a standard protocol for participants with chronic pain and insomnia.

Objective: To assess the feasibility and acceptability of AA and to evaluate the effectiveness of AA on pain severity score, pain interference score, and insomnia over an 8-day study period.

Subjects: 45 participants who met the eligibility criteria and signed the consent were randomized to either the AA group (AAG) or the usual care control group (CG) on day 4.

Intervention: A standard AA protocol using penetrating semi-permanent acupuncture needles and in-place for up to four days.

Main Outcome Measures: Brief Pain Inventory pain severity and interference scores for pain and Insomnia Severity Index (ISI) for insomnia.

Results: The use of the standard AA protocol in the AAG led to significant within- and between-group reduction in pain severity and interference scores when compared to the CG. Both groups showed within-group decrease in ISI. However, the AAG showed significant between-group reduction in ISI severity and from moderate to sub-threshold insomnia.

Conclusions: AA was found to show effectiveness in the treatment of chronic pain and insomnia. With a heightened focus on the opioid crisis in the U.S., this easy-to-administer protocol can be an option for treatment modality for military beneficiaries with chronic pain and insomnia.

ELIGIBILITY:
Inclusion Criteria:

* military beneficiary - active duty, retiree, or dependents
* between the ages of 18 - 65 years
* fall under the care of LRMC footprint
* self-report of insomnia based on established research criteria
* sleep-onset latency (SOL) or wakefulness after sleep onset of ≥30 minutes;

  * frequency of at least three times a week;
  * duration of ≥3 months;
  * with unrestorative or unrefreshing sleep
* NRS Pain rating ≥3 (mild to severe level)
* pain for ≥3 months
* able to read and understand English
* for active duty military, an agreement of supervisor

Exclusion Criteria:

* hypersensitivity or allergy to gold.
* pregnancy or plan for future pregnancy during the duration of the study (since the safety of AA in pregnant women has not been established; based on self-report rather than requiring a pregnancy test)
* ear trauma or unhealed wounds on the ear
* participation in any other research protocol with a device or drugs
* piercing or scar tissue in any of the AA point areas
* working in jobs with variable hours (e.g., shift work)
* acupuncture treatment within the last 3 months
* individuals with valvular prosthetics, hemophilia, or currently receiving an anticoagulant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index over time | Baseline, day 4, day 8
  Insomnia Severity Index (ISI). Assesses the perceived severity and impact of insomnia symptoms based on a 5-point Likert with a total score from 0-28 with >14 indicating moderate to severe insomnia. The sensitivity and specificity are 94% using a cutoff score of 14. Good test-retest (.78), face validity as defined by DSM-IV, and concurrent validity (.32 - .99)

SECONDARY OUTCOMES:
Change in Sleep Diary components over time | Daily for duration of study
  Sleep Diary 69. Collects and quantifies daily, subjective bedtime and waketime sleep parameters 70. A sleep diary in various formats is often used as a diagnostic tool for sleep disorders. In addition, due to one major weakness of validity check of real time completion, the sleep diary is often used in conjunction with actigraphy to establish validity in sleep parameters. Based on the recommendations for standard research assessment, a sleep diary should assess the following information: sleep onset latency (SOL), final waketime, number of awakenings (NWAK), wake after sleep onset (WASO), total sleep time (TST), sleep efficiency (SE), sleep quality (SQ), and time/duration of naps. Sleep diaries are standard practice and recommended for use in research studies of sleep disorder treatments.
Change in Actigraphy measures over time | Daily for duration of study
  Actigraphy is a watch-like device that documents sleep/wake patterns via movement over a period of time to estimate sleep parameters. It records in-time blocks (epochs) the participant's movement, light exposure, and other measures using accelerometry and a light meter. Various clinical research studies that have compared the outcomes among actigraphy vs. polysomnography (PSG) - the gold standard in sleep research. Correlation rates have been >90% in healthy adults and >84% in patients with sleep related breathing disorders when actigraphy has been compared to PSG 73,74. For Actiwatch 2, scoring software of Actiware will be used to determine sleep parameters of SOL, NWAK, WASO, TST, and SE.
Change in Brief Pain Inventory over time | Daily for duration of Study
  . Assesses four pain items and the degree of interference with seven aspects of functioning using a 0-10 Numeric Rating Scale. Four pain items include "pain now," "pain at its worst," "pain at its least," and "average" over the last 24 hours. The BPI also includes the location of pain on a body chart and the use of pain medications. "Worst pain" or the arithmetic mean of the 4 severity items can be used as measures of pain severity and the arithmetic mean of the 7 interference items can be used a as a measure of pain interference. Validity and reliability are high in various chronic pain populations (.77-.91)
Change in Defense and Veterans Pain Scale over time | Daily for duration of Study
  This 5-item scale was developed by a 22-member Pain Management Task Force as a standard pain assessment in the Department of Defense (DoD)/Veterans Administration (VA) system for continuity of care of service members. However, there are very few studies on its validity and reliability. The scale integrates a currently used numeric pain rating scale with visual facial cues and word descriptors. In addition there are 4 supplemental questions on pain interference modified from the BPI. Construct validity using component factor analysis revealed one item group (factor loadings >.78 and >.81) for outpatient and inpatient participants, respectively, with high internal consistency (.87-.90)

CONTACTS AND LOCATIONS:
Overall Officials: Ann K Ketz, PhD, Principal Investigator — Landstuhl Regional Medical Center
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, APO AE, Germany

IPD SHARING:
Plan to Share IPD: Undecided